CLINICAL TRIAL: NCT00035074
Title: A Pharmacokinetic Study to Determine the Oral Bioavailability of Methotrexate in Patients With Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Crohn's and Colitis Foundation (Other)
Model: Crossover | Purpose: Treatment
Other Study IDs: NCRR-M01RR00240-1757
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Methotrexate

INTERVENTIONS:
Drug: Methotrexate

SUMMARY:
Patients with inflammatory bowel disease (IBD) who require methotrexate (MTX)for treatment currently receive this drug by injection. MTX is also available as a pill that can be given by mouth but it is not known how well the drug enters the body in patients with Crohn's disease or ulcerative colitis. This study is being done to compare how much MTX enters the body when the drug is taken by mouth compared to when it is given by injection. If the drug is well absorbed, it may allow patients to receive the drug by mouth.

ELIGIBILITY:
* Adult or pediatric patients with IBD (CD or UC) currently receiving MTX as part of their clinical care.
* Patients must be receiving weekly MTX at a dose between 7.5 and 40 mg/m2.
* Weight >= 12 kg.
* Normal serum creatinine.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania, United States